CLINICAL TRIAL: NCT05277753
Title: NGS-MRD Evaluation of Antigen-specific T Cells and DC Vaccine Combination Targeting T-cell Acute Lymphoblastic Leukemia
Brief Title: NGS-MRD Assessment of Combination Immunotherapies Targeting T-ALL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-22002
Record Dates: First submitted 2022-02-21; First posted 2022-03-14 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: T-Cell Acute Lymphoblastic Leukemia
Keywords: T-ALL; CAR T; CTL; DC vaccine
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — S-1,2-dichlorovinyl-N-acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CART/CTL/DCvac cells to treat T-ALL (Experimental)
  Interventions: Biological: Antigen-specific T cells CAR-T/CTL and DCvac

INTERVENTIONS:
Biological: Antigen-specific T cells CAR-T/CTL and DCvac — Antigen-specific T cells CAR-T/CTL and DCvac cells to treat T-ALL

SUMMARY:
The purpose of this study is to determine the feasibility, safety, and efficacy of a combination therapy in the treatment of T-cell acute lymphoblastic leukemia (T-ALL): multi-antigen-targeted chimeric antigen receptor T cells (CAR-T) followed by engineered immune effector cytotoxic T cells (CTLs) and immune modified dendritic cell vaccine (DCvac). This approach is aimed to achieve NGS MRD negativity in T-ALL patients, which can identify a very low risk of relapse and define patients with possible long-term remission without further treatment.

DETAILED DESCRIPTION:
Minimal residual disease (MRD) monitoring is currently performed in T-ALL patients to evaluate treatment response and define risk stratification. Patients with good prognosis have undetectable MRD levels after treatment, while persistent MRD defines high relapse-risk patients. The standardized flow cytometry assay detects MRD reliably in bone marrow or peripheral blood at levels ≥0.01% mononuclear cells. More sensitive MRD assay detecting specific clonal T cell receptors (TCR) by next-generation sequencing (NGS) can reliably detect blasts at levels ≤10-6 cells. Given the high sensitivity, NGS-MRD approach improves distinction between deeply negative and very low positive cases. Recent studies also demonstrate that NGS-MRD assessment of the bone marrow with undetectable blast cells is a strong predictive factor, indicating patients with possible long-term response after CAR-T cell therapy.

Acute lymphoblastic leukemia (ALL) is hematological malignancy with the highest incidence in children and adolescents. After standardized treatment, the survival rate is relatively high. ALL is divided into two types: B cells and T cells, the latter accounting for about 15% of childhood leukemias and about 25% of adult leukemias. Compared with children and adolescents with B-lineage ALL (B-ALL), T-ALL is extremely aggressive, and patients are prone to early disease recurrence, and in the event of recurrence, event-free survival (EFS) and overall survival (OS) are lower, at less than 25%, even with more intensive treatment, which might require further combination therapy to enhance anti-tumor immunity and eradicate all malignant cells. Therefore, this protocol includes multi-target CAR-T cell infusions followed by antigen-specific cytotoxic T lymphocyte (CTL)-based immunotherapy, which is based on T cells reacting with specific T-ALL tumor antigens and immune-modified dendritic cells (DCvac) fused with T leukemic cells as DC vaccines. In addition to the significant success of CAR-T cell therapy, various clinical studies also reported the importance and potential benefits of using tumor-specific T cells in different types of cancer. Moreover, DC-based vaccines as another agent of immunotherapy have proven to prevent or delay relapse in leukemia patients achieving remission. In this study, we combine those strategies to augment anti-tumor immunity in patients and expect undetectable NGS-MRD, a long-lasting remission to prevent disease recurrence.

We propose a novel protocol which combines multi-CAR-T cell therapy, engineered immune effector CTLs and DCvac against T-ALL. The aim of this study is to evaluate the feasibility, safety, and efficacy of the NGS-MRD analysis-based combinational immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 6 months.
2. High-burden (≥ 30% blast cells) bone marrow sample for NGS TCR clonal identification and CTL/DC vac preparation is required
3. Expression of CD7, CD5, CD317, CD47, CD99, CD38 or TRBC1/2 is determined in malignant cells by flow cytometry or immuno-histochemical staining.
4. Karnofsky performance status (KPS) score is higher than 80 and life expectancy > 3 months.
5. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: cardiac ejection fraction ≥ 50%, oxygen saturation ≥ 90%, creatinine ≤ 2.5x upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3x upper limit of normal, total bilirubin ≤ 2.0 mg/dL.
6. Hgb ≥ 80g/L.
7. No cell separation contraindications.
8. Abilities to understand and the willingness to provide written informed consent.

Exclusion Criteria:

1. Sever illness or medical condition, which would not permit the patient to be managed according to the protocol, including active uncontrolled infection.
2. Active bacterial, fungal or viral infection not controlled by adequate treatment.
3. Known HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
4. Pregnant or nursing women may not participate.
5. History of glucocorticoid for systemic therapy within the week prior to entering the test.
6. Previous treatment with any gene therapy products.
7. Patients, in the opinion of investigators, may not be eligible or not able to comply with the study.

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-related adverse events are assessed by NCI CTCAE V4.0 criteria. | 1 year
  Safety of infusion
Clinical response | 1 year
  Leukemia blast cells are detected by multiparameter flow cytometry
Evaluate the percentage of minimal leukemia residue in bone marrow | 1 year
  Minimal leukemia residue（MRD）is measured by TCR next generation sequencing（NGS）.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China